CLINICAL TRIAL: NCT06573398
Title: Efficacy and Safety of Radiotherapy With Sequential Chemotherapy Combined With PD-1 Inhibitor and Thymalfasin for Borderline Resectable Pancreatic Cancer
Brief Title: Radiotherapy With Sequential Chemotherapy Combined With PD-1 Inhibitor and Thymalfasin for BRPC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, JIABIN JIN, Associate Chief Physician, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDX+PD-1+CRT-PDAC
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: borderline resectable; thymalfasin; radiotherapy; chemotherapy; PD-1 inhibitor; pancreatic ductal adenocarcinoma
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRT+PD-1 inhibitor+Thymalfasin (Experimental): All eligible 20 subjects will receive a neoadjuvant therapy regimen of chemoradiotherapy combined with anti-PD-1 monoclonal antibody and Thymalfasin.
  Interventions: Combination Product: SBRT with Sequential AG regimen +Tislelizumab+Thymalfasin

INTERVENTIONS:
Combination Product: SBRT with Sequential AG regimen +Tislelizumab+Thymalfasin — Stereotactic body radiation therapy (SBRT): 30 ~ 40 Gy/5f, Week 1, Day 1 ~ Day 5, 6-8 Gy/time, once a day; 3 weeks as a cycle, for 4 cycles Tislelizumab: 200 mg, i.v., single infusion, 21 days as a cycle for 4 cycles, on Day 1 of each treatment cycle; Thymalfasin: 4.8 mg, subcutaneous injection, twice a week, on Day 1 and Day 4 of each week during Weeks 1 ~ 13; Albumin-bound paclitaxel: 125 mg/m2, i.v., on Day 1 and Day 8 of each treatment cycle; Gemcitabine: 1000mg/m2, i.v., on Day 1 and Day 8 of each treatment cycle; After 4 cycles of preoperative neoadjuvant therapy, radical surgery will be evaluated by the MDT team within 2-4 weeks after completion of chemotherapy + immunotherapy.

SUMMARY:
This is a prospective, single-center, single-arm, phase II clinical study. The primary purpose of the study was to evaluate the efficacy and safety of radiotherapy with sequential albumin-bound paclitaxel + Gemcitabine chemotherapy + anti-PD-1 monoclonal antibody and Thymalfasin for borderline resectable pancreatic cancer, and to explore clinical indicators related to efficacy, further guiding subsequent individualized precise treatment.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm, phase II clinical study. In this study, 20 patients with borderline resectable pancreatic cancer and without any prior treatment will be enrolled. After signing the informed consent form, patients will be screened to ensure they meet the eligibility criteria.Before surgery, eligible patients will receive 4 cycles of neoadjuvant therapy: Tislelizumab combined with AG regimen and SBRT and 13 weeks of Thymalfasin therapy; after 4 cycles, the efficacy will be evaluated and radical surgery will be performed on schedule. The postoperative treatment of patients will be jointly decided by clinical physicians and patients according to the actual conditions of clinical diagnosis and treatment.

The main observation indicator is the R0 resection rate after neoadjuvant therapy; Safety assessment: The safety will be assessed after each cycle of neoadjuvant therapy and at 30 days after the last dose; Event follow-up: The events will be followed once every 3 months during the first year after surgery, and once every 6 months during the second year after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, with ECOG score of 0 ~ 1;
2. Histologically or cytologically confirmed diagnosis of ductal adenocarcinoma of pancreas;
3. Classification as borderline resectable pancreatic cancer according to the NCCN Guidelines (2024 Edition);
4. Deemed suitable for neoadjuvant therapy following discussion by the MDT team of the study site;
5. Subjects must meet the following criteria for hematology test:

   1. Neutrophil count ≥ 1.5 × 10^9/L
   2. Hemoglobin ≥ 10 g/dL
   3. Platelet count ≥ 100 × 10^9/L
6. Subjects must meet the following criteria for blood chemistry tests:

   1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   2. AST and ALT < 1.5 × ULN
   3. Creatinine clearance ≥ 60 mL/min
   4. Good coagulation, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN
7. Subjects of childbearing potential should take appropriate protective measures (contraceptive methods or other birth control methods) prior to enrollment and throughout the clinical study;
8. Has signed the informed consent form;
9. Capable of complying with the study protocol and follow-up procedures.

Exclusion Criteria:

1. Prior systemic anti-tumor therapy;
2. Prior medical history of other tumors, except for cervical carcinoma in situ, treated squamous cell carcinoma or urothelial bladder carcinoma (Ta and TIS), or other malignant tumors that have received radical treatment (at least 5 years prior to enrollment);
3. Prior history of abdominal radiotherapy;
4. Subjects with active bacterial or fungal infection (≥ Grade 2 as per NCI-CTC, Version 3).
5. Subjects with HIV, HCV, or HBV infection, uncontrollable coronary artery disease or asthma, uncontrollable cerebrovascular disease or other diseases judged by the investigator to be ineligible for enrollment;
6. Subjects with autoimmune diseases or immunodeficiency and requiring treatment with immunosuppressive agents;
7. Pregnant or lactating women; women of childbearing potential must have a negative pregnancy test results within 7 days prior to enrollment;
8. Subjects with drug abuse/clinical/psychological/social factors that affect informed consent or study conduct;
9. Subjects who may be allergic to PD-1 monoclonal antibody immunotherapy drugs;
10. Patients who are scheduled to undergo or have previously undergone organ or bone marrow transplant;
11. Patients requiring treatment with systemic corticosteroids (at dose level > 10 mg/day prednisone efficacy) or other immunosuppressive drugs within 14 days prior to the first dose or during the study. However, enrollment is permitted if: In the absence of active autoimmune disease, patients are permitted to use topical or inhaled steroids, or adrenal hormone replacement therapy at dose level ≤ 10 mg/day prednisone efficacy;
12. Treatment with live vaccines within 28 days prior to the first dose; except for inactivated viral vaccines for seasonal influenza;
13. Active pulmonary tuberculosis;
14. Treatment with related drugs or medical technology affecting immunity within 6 months prior to the first dose (including but not limited to: thymopentin, thymalfasin, interferon, CAR-T therapy, etc.);
15. Patients with other conditions unsuitable for this clinical trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | within 10 days after surgery
  Defined as the proportion of patients in the ITT population who undergo R0 resection following neoadjuvant therapy among patients undergoing surgery.

SECONDARY OUTCOMES:
Tumor regression grade (TRG) | within 10 days after surgery
  Tumor regression grade was determined according to the postoperative pathological results.
Pathologic complete response (pCR) rate | within 10 days after surgery
  Defined as the proportion of patients in the ITT population who reach pT0N0M0 among patients undergoing surgery.
Median progression-free survival (mPFS) | 24 months
  The median time from the first dose to any documented tumor progression or death due to any cause (whichever occurs first) in the ITT population. Patients who are alive at the time of analysis and have no documented disease progression will be reviewed on the date of the last imaging assessment.
Median overall survival (mOS) | 24 months
  The median time from the first dose to death due to any cause in the ITT population. Patients who are alive at the time of analysis will be reviewed on their last contact date.
Major pathologic response (MPR) rate | within 10 days after surgery
  Defined as the proportion of patients in the ITT population who achieve TRG1 among patients undergoing surgery.
Objective response rate (ORR) | Baseline (before surgery)
  Defined as the proportion of patients in the ITT population achieving complete response (CR) + partial response (PR) according to iRECIST.
Disease control rate (DCR) | Baseline (before surgery)
  Defined as the proportion of subjects in the ITT population who achieve disease response and stable disease among all subjects.
TRAE | from commencing of treatment to the 30th day after surgery
  Incidence of treatment-related adverse event
irAE | from commencing of PD-1 inhibitor to the 30th day after surgery
  Incidence of immune-related adverse event
Incidence of surgical complications | within 30 days after surgery
  Incidence of surgical complications within 30 days after surgery

OTHER OUTCOMES:
The expression of CD68 | up to 3 months after surgery
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC
The expression of CD86 | up to 3 months after surgery
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC
The expression of CD163 | up to 3 months after surgery
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC
The expression of CD4 | up to 3 months after surgery
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC
The expression of CD8 | up to 3 months after surgery
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC

CONTACTS AND LOCATIONS:
Overall Officials: Baiyong Shen, PhD,MD, Principal Investigator — Ruijin Hospital; Jiabin Jin, PhD, Principal Investigator — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No
Export of individual patient data is a sensitive issue according to current Chinese laws.